CLINICAL TRIAL: NCT02412826
Title: Abstats: Computer-aided, Non-invasive, Acoustic Gastrointestinal Surveillance (AGIS) in Acute Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Elham Afghani, Assistant Director, Clinical Pancreatology, Cedars-Sinai Medical Center
Other Study IDs: Pro00038455
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Pancreatitis
Keywords: pancreatitis; acoustic; sensor
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute pancreatitis: Patients presenting to the hospital with acute pancreatitis that will receive AbStats sensor
  Interventions: Device: Abstats sensor

INTERVENTIONS:
Device: Abstats sensor — The AbStats abdominal biosensor will be applied to the abdomen of patients who are admitted with acute pancreatitis.

SUMMARY:
The purpose of this study is to conduct a pilot test of an abdominal acoustic sensor on patients with acute pancreatitis to determine the correlation of acoustic signals with symptoms reported by the patient.

DETAILED DESCRIPTION:
This study will use the AbStats device, that measure IAAS (intraabdominal acoustic signals) and intestinal rate and will correlate this data with symptoms reported by patients hospitalized for acute pancreatitis.

The AbStats multi-sensor wireless abdominal monitoring system includes low profile acoustic sensors that are applied to the anterior abdominal wall with Tegaderm and monitors sounds emanating from the GI tract. The acoustic sensors continuously and non-invasively monitor and capture audio signals representing GI and abdominal wall function. The captured data is recorded in a synchronized manner from all sensors.

We will place the AbStats sensor on all patients immediately after admission to the hospital. Only study staff trained on the AbStats system will apply the sensors, which fit externally around the abdomen. A physician member of our study staff will be available at all times to help position the device if needed. We will continuously record AbStats acoustic signals for the duration of the hospitalization, with the option to discontinue as clinically required or requested by the provider or patient. A research coordinator will collect clinical data from medical records and enter the data into a secure spreadsheet on CSMC servers. Patients will be asked to keep a daily diary of symptoms. In this diary, the patients will be asked to record information about their food consumption (if any), bowel movements (if any and if associated with contrast from CT imaging or with the use of suppositories/ laxative), specific symptoms, and whether the sensor was removed for any period of time during the day. This will allow us to compare the data collected by the AbStats sensor with self-reported symptoms noted by patients. Physicians and nurses will not be made aware of the AbStats readings so as to eliminate the Hawthorne effect. Patients will be managed according to standard-of-care practice and the data collected by the AbStats device will not be incorporated into clinical care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* diagnosis of acute pancreatitis; must meet at least 2 out of the 3 following critiera:

  1. abdominal pain consistent with acute pancreatitis
  2. serum amylase/lipase >3 times upper limit of normal
  3. characteristic findings from abdominal imaging
* able to provide informed consent

Exclusion Criteria:

* unable to provide consent
* transfer patients
* cognitive inability to follow directions to maintain sensors in place
* unable to place abdominal sensors on patients
* abdominal cellulitis
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients who present to Cedars-Sinai Medical Center with the diagnosis of acute pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Re-hospitalization for acute pancreatitis | 30 days
  Patients who are re-admitted to the hospital for acute pancreatitis
Ability to PO after discharge | 30 days
  Patients who are able to tolerate oral itnake after discharge
Symptoms | 30 days
  GI symptoms after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Elham Afghani, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Negro P, D'Amore L, Saputelli A, Talarico C, Scaccia M, Tuscano D, Gossetti F, Carboni M. Colonic lesions in pancreatitis. Ann Ital Chir. 1995 Mar-Apr;66(2):223-31. PMID 7668499
- [Background] Abcarian H, Eftaiha M, Kraft AR, Nyhus LM. Colonic complications of acute pancreatitis. Arch Surg. 1979 Sep;114(9):995-1001. doi: 10.1001/archsurg.1979.01370330017003. PMID 485850
- [Background] Russell JC, Welch JP, Clark DG. Colonic complications of acute pancreatitis and pancreatic abscess. Am J Surg. 1983 Nov;146(5):558-64. doi: 10.1016/0002-9610(83)90288-x. PMID 6638261
- [Background] Shi LL, Liu MD, Chen M, Zou XP. Involvement of interstitial cells of Cajal in experimental severe acute pancreatitis in rats. World J Gastroenterol. 2013;19(14):2179-86. doi: 10.3748/wjg.v19.i14.2179. PMID 23599644
- [Background] Leveau P, Wang X, Soltesz V, Ihse I, Andersson R. Alterations in intestinal motility and microflora in experimental acute pancreatitis. Int J Pancreatol. 1996 Oct;20(2):119-25. doi: 10.1007/BF02825510. PMID 8968867
- [Background] Seerden TC, De Man JG, Holzer P, Van den Bossche RM, Herman AG, Pelckmans PA, De Winter BY. Experimental pancreatitis disturbs gastrointestinal and colonic motility in mice: effect of the prokinetic agent tegaserod. Neurogastroenterol Motil. 2007 Oct;19(10):856-64. doi: 10.1111/j.1365-2982.2007.00968.x. PMID 17883437
- [Background] Wang X, Gong Z, Wu K, Wang B, Yuang Y. Gastrointestinal dysmotility in patients with acute pancreatitis. J Gastroenterol Hepatol. 2003 Jan;18(1):57-62. doi: 10.1046/j.1440-1746.2003.02898.x. PMID 12519225
- [Background] Davis S, Parbhoo SP, Gibson MJ. The plain abdominal radiograph in acute pancreatitis. Clin Radiol. 1980 Jan;31(1):87-93. doi: 10.1016/s0009-9260(80)80088-2. PMID 7357829
- [Background] Asgeirsson T, El-Badawi KI, Mahmood A, Barletta J, Luchtefeld M, Senagore AJ. Postoperative ileus: it costs more than you expect. J Am Coll Surg. 2010 Feb;210(2):228-31. doi: 10.1016/j.jamcollsurg.2009.09.028. Epub 2009 Nov 18. PMID 20113944
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Background] Yadav D, Lee E, Papachristou GI, O'Connell M. A population-based evaluation of readmissions after first hospitalization for acute pancreatitis. Pancreas. 2014 May;43(4):630-7. doi: 10.1097/MPA.0000000000000078. PMID 24681876
- [Background] Vipperla K, Papachristou GI, Easler J, Muddana V, Slivka A, Whitcomb DC, Yadav D. Risk of and factors associated with readmission after a sentinel attack of acute pancreatitis. Clin Gastroenterol Hepatol. 2014 Nov;12(11):1911-9. doi: 10.1016/j.cgh.2014.04.035. Epub 2014 May 9. PMID 24815327
- [Background] Tomomasa T, Morikawa A, Sandler RH, Mansy HA, Koneko H, Masahiko T, Hyman PE, Itoh Z. Gastrointestinal sounds and migrating motor complex in fasted humans. Am J Gastroenterol. 1999 Feb;94(2):374-81. doi: 10.1111/j.1572-0241.1999.00862.x. PMID 10022632
- [Background] Augustyniak P. Wearable wireless heart rate monitor for continuous long-term variability studies. J Electrocardiol. 2011 Mar-Apr;44(2):195-200. doi: 10.1016/j.jelectrocard.2010.11.014. PMID 21353066
- [Background] Shambroom JR, Fabregas SE, Johnstone J. Validation of an automated wireless system to monitor sleep in healthy adults. J Sleep Res. 2012 Apr;21(2):221-30. doi: 10.1111/j.1365-2869.2011.00944.x. Epub 2011 Aug 22. PMID 21859438
- [Background] Spiegel BM, Kaneshiro M, Russell MM, Lin A, Patel A, Tashjian VC, Zegarski V, Singh D, Cohen SE, Reid MW, Whitman CB, Talley J, Martinez BM, Kaiser W. Validation of an acoustic gastrointestinal surveillance biosensor for postoperative ileus. J Gastrointest Surg. 2014 Oct;18(10):1795-803. doi: 10.1007/s11605-014-2597-y. Epub 2014 Aug 5. PMID 25091837